CLINICAL TRIAL: NCT00827190
Title: Ascending Single Dose Study Of The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of ILS-920 Administered Intravenously To Healthy Adult Subjects
Brief Title: Study Evaluating Single Ascending Doses Of ILS-920
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3216K1-1000
Record Dates: First submitted 2008-12-10; First posted 2009-01-22 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-02

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): ILS-920
  Interventions: Drug: ILS-920

INTERVENTIONS:
Drug: ILS-920

SUMMARY:
This is a first-in-human study of ILS-920. This study will provide an initial assessment of the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of ILS-920 after administration of ascending single intravenous (IV) doses to healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men or women of nonchildbearing potential
* Aged 18 to 50 years inclusive at screening.

Exclusion Criteria:

* Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
* History of drug abuse within 1 year before study day 1.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Safety based on vital sign evaluations, 12-lead ECGs, cardiac rhythm monitoring and routine lab tests. | 48 hours after study drug administration

SECONDARY OUTCOMES:
Pharmacokinetics will measure the extent and rate of Absorption, Distribution, Metabolism and Excretion of the drug in the body. | 48 hours after study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer